CLINICAL TRIAL: NCT01124812
Title: A Prospective Non-randomized Study of 131I-L19SIP Radioimmunotherapy (RIT) in Combination With External Beam Radiotherapy (EBRT) and Concurrent Chemotherapy in Patients With Inoperable, Locally-advanced (Stage III) NSCLC
Brief Title: 131I-L19SIP Radioimmunotherapy Combined With Radiochemotherapy in Patients With Locally-advanced Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19SIPI131-04/09; 2009-017072-24 (EudraCT Number)
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: I131; L19; antibody; monoclonal; NSCLC; lung; tumor targeting; radioimmunotherapy; Patients with newly diagnosed inoperable, locally-advanced (stage III) NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 131I-L19SIP (Experimental): 131I-L19SIP Radioimmunotherapy (RIT) in Combination With External Beam Radiotherapy (EBRT) and Concurrent Chemotherapy: Treatment dose of 131I-L19SIP RIT is titrated in cohorts of 3 patients.
  Interventions: Other: 131I-L19SIP Radioimmunotherapy (RIT) in Combination With External Beam Radiotherapy (EBRT) and Concurrent Chemotherapy

INTERVENTIONS:
Other: 131I-L19SIP Radioimmunotherapy (RIT) in Combination With External Beam Radiotherapy (EBRT) and Concurrent Chemotherapy — Lung tumor irradiation with a total dosage of between 60-66 Gy, fractionated in combination with the following concurrent chemotherapy options:
  1. Cohorts 1, 2 & 3a is composed of cisplatin i.v. 80 mg/m2 on day 1, and vinorelbine i.v. 25 mg/m2 on day 1, 8, 15 for cycle 1 & 4. For patients with significant comorbidities, the dose of vinorelbine is reduced to 12.5 mg/m2 during cycles 2 & 3. Treatment cycles will be repeated every 28 days.
  2. Protocol A (suggested for patients with comorbidities: Carboplatin 70 mg/m2, over 30 min iv, (Day 1-5 ) + Vinorelbine 12.5 mg/m2 as a 5-min bolus iv or short iv-infusion (Day 1, 8, 22), repeated on Day 28.
  3. Protocol B (suggested for patients in good clinical condition): Paclitaxel 50 mg/m2 1 hour iv (Day 1, 15, 22, 29, 36, 43, 50) + Carboplatin AUC 2, 30 min iv on (Day 1, 15, 22, 29, 36, 43, 50).
     * Total treatment duration is 8-16 weeks

SUMMARY:
The aim of this feasibility study is to determine the therapeutic potential of the L19SIP antibody, labeled with the radionuclide 131I in combination with radiochemotherapy, for the treatment of patients with newly diagnosed, unresectable, locally-advanced NSCLC following the promising results with this agent in previous clinical studies.

The L19SIP antibody is a fully human antibody, capable of preferential localization around tumor blood vessels while sparing normal tissues. The formation of new blood vessels is a rare event in the adult (with the exception of the female reproductive tract), but it is a characteristic pathological feature for most types of aggressive cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable stage III NSCLC
* Males or females, age ≥ 18 years
* Measurable lung lesion defined as at least one lesion that can be accurately and serially measured per the modified RECIST criteria.
* ECOG performance status < 3
* Life expectancy of at least 12 weeks
* Patients eligible for concurrent radiochemotherapy (cisplatin/vinorelbine; 60-66 Gy EBRT) at the discretion of the clinical investigator
* Absolute neutrophil count > 1.5 x 109/L, hemoglobin > 9.0 g/dL and platelets > 100 x 109/L
* Total bilirubin ≤ 30 µmol/L (or ≤ 2.0 mg/Dl)
* ALT and AST ≤ 2.5 x the upper limit of normal (5.0 x ULN for patients with hepatic involvement with tumor
* Serum creatinine < 1.5 x ULN
* All toxic effects of prior therapy must have resolved to ≤ Grade 1 unless otherwise specified above
* Negative serum pregnancy test (for women of child-bearing potential only) at screening

Exclusion Criteria:

* Patients with metastatic disease
* Patients amenable for surgical resection of lung tumor lesions
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, Tis & Ti) or any cancer curatively treated < 5 years prior to study entry
* History of HIV infection or infectious hepatitis B or C
* Presence of active infections (e.g. requiring antibimicrobial therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Inadequately controlled cardiac arrhythmias including atrial fibrillation
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria)
* Uncontrolled hypertension
* Ischemic peripheral vascular disease (Grade IIb-IV)
* History of an acute cardiac event such as myocardial infarction, instable angina pectoris during the last 12 months
* Severe diabetic retinopathy
* Active autoimmune disease
* History of organ allograft or stem cell transplantation
* Recovery from major trauma including surgery within 4 weeks prior to administration of study treatment
* Breast feeding female
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment
* Growth factors or immunomodulatory agents within 7 days of the administration of study treatment (131I-L19SIP application).
* Hyperthyroidism or autonomous thyroid nodule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Uptake of 131I-L19SIP or 124I-L19SIP | 2 days
  The selective uptake of 131I-L19SIP or 124I-L19SIP in lung lesions and dosimetric analysis
Safety and tolerability of 131I-L19SIP Radioimmunotherapy (RIT) in Combination With External Beam Radiotherapy (EBRT) and Concurrent Chemotherapy | 13 months
  Safety will be assessed through physical examinations, vital signs, laboratory tests (including serum chemistries, hematology parameters) and the recording of adverse events. All results from these assessments will be coded using CTCAE v.3 and presented descriptively, indicating frequency and percentage of patients with adverse events, and abnormal laboratory tests. These results will be presented by related/unrelated and overall for the study.
Dose Limiting Toxicities (DLTs) and Maximum Tolerated Dose/Recommended Dose (MTD/RD) for the combination treatment | 4 weeks
  Dose limiting toxicities and maximum tolerated dose/recommended dose for the combination treatment

SECONDARY OUTCOMES:
Overall response rate | 1 year
  Intrapulmonal, extra pulmonal and overall response rate
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Paganelli, Dr, Principal Investigator — IRST - ISTITUTO SCIENTIFICO ROMAGNOLO PER LO STUDIO E LA CURA DEI TUMORI - MELDOLA (FC)
Locations (2):
- Italy (2):
  - University Hospital Pisa, Pisa, Tuscany
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Meldola (Fc), Meldola